CLINICAL TRIAL: NCT00654381
Title: A Double-blind Phase III Study to Evaluate the Efficacy of BI 1356 5 mg and 10 mg vs. Placebo for 12 Weeks and vs. Voglibose 0.6 mg for 26 Weeks in Patients With Type 2 Diabetes Mellitus and Insufficient Glycaemic Control, Followed by an Extension Study to 52 Weeks to Evaluate Long-term Safety
Brief Title: Japanese P III vs Voglibose and Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.23
Record Dates: First submitted 2008-04-03; First posted 2008-04-08 (Estimated); Results first posted 2011-08-02 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; voglibose

ARMS (4):
- voglibose 0.2 mg three times a day (TID) (Active Comparator): patient to receive a tablet containing 0.2 mg voglibose TID plus 2 placebo tablets matching BI 1356
  Interventions: Drug: voglibose
- BI 1356 low dose (Experimental): patient to receive a tablet containing BI 1356 and matching placebo plus 3 placebo tablets matching voglibose
  Interventions: Drug: BI 1356
- BI 1356 high dose (Experimental): patient to receive 2 tablets containing BI 1356 plus 3 placebo tablets matching voglibose
  Interventions: Drug: BI 1356
- placebo (Placebo Comparator): patient to receive 2 placebo tablets matching BI 1356 plus 3 placebo tablets matching voglibose
  Interventions: Drug: voglibose placebo; Drug: BI 1356 placebo

INTERVENTIONS:
Drug: BI 1356 — 5 mg/daily
  Arms: BI 1356 low dose
Drug: BI 1356 — 10 mg/daily
  Arms: BI 1356 high dose
Drug: voglibose placebo — three times daily
  Arms: placebo
Drug: BI 1356 placebo — once daily
  Arms: placebo
Drug: voglibose — 0.6 mg/daily
  Arms: voglibose 0.2 mg three times a day (TID)

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and tolerability of Linagliptin (BI 1356) (5 mg or 10 mg / once daily) compared to placebo given for 12 weeks and voglibose for 26 weeks as mono therapy in patients with type 2 diabetes mellitus with insufficient glycaemic control. Furthermore, long-term safety is evaluated with an extension treatment to 52 weeks.

ELIGIBILITY:
Inclusion criteria:

1. Japanese patients with a diagnosis of type 2 diabetes mellitus. Antidiabetic therapy has to be stable for at least 10 weeks before Visit 1.
2. Glycosylated haemoglobin A1 (HbA1c) 7.0 - 10.0% at Visit 3 (beginning of the 2-week placebo run-in phase)
3. Age: >= 20 and <= 80
4. Body Mass Index (BMI) <= 40 kg/m2

Exclusion criteria:

1. Myocardial infarction, stroke or transient ischemic attack (TIA) within 6 months before Visit 1
2. Impaired hepatic function
3. History of severe allergy/hypersensitivity
4. Treatment with anti-diabetic, anti obesity drugs, etc 3 months before Visit 1
5. Fasting blood glucose >240 mg/dl (=13.3 mmol/L) at Visits 2 or 3

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2008-04; Primary Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (47):
- Japan (47):
  - 1218.23.05 Boehringer Ingelheim Investigational Site, Asahi, Chiba
  - 1218.23.06 Boehringer Ingelheim Investigational Site, Funabashi, Chiba
  - 1218.23.21 Boehringer Ingelheim Investigational Site, Hitachinaka, Ibaraki
  - 1218.23.44 Boehringer Ingelheim Investigational Site, Hitachiota, Ibaraki
  - 1218.23.09 Boehringer Ingelheim Investigational Site, Imizu, Toyama
  - 1218.23.45 Boehringer Ingelheim Investigational Site, Inashiki-gun, Ibaraki
  - 1218.23.13 Boehringer Ingelheim Investigational Site, Izumisano, Osaka
  - 1218.23.27 Boehringer Ingelheim Investigational Site, Kariya, Aichi
  - 1218.23.47 Boehringer Ingelheim Investigational Site, Kitakatsushika-gun, Saitama
  - 1218.23.39 Boehringer Ingelheim Investigational Site, Kitakyuushuu, Fukuoka
  - 1218.23.02 Boehringer Ingelheim Investigational Site, Koriyama, Fukushima
  - 1218.23.03 Boehringer Ingelheim Investigational Site, Koriyama, Fukushima
  - 1218.23.10 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 1218.23.37 Boehringer Ingelheim Investigational Site, Marugame, Kagawa
  - 1218.23.38 Boehringer Ingelheim Investigational Site, Marugame, Kagawa
  - 1218.23.23 Boehringer Ingelheim Investigational Site, Matsumoto, Nagano
  - 1218.23.07 Boehringer Ingelheim Investigational Site, Meguro-ku, Tokyo
  - 1218.23.25 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1218.23.26 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1218.23.28 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1218.23.29 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1218.23.30 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1218.23.04 Boehringer Ingelheim Investigational Site, Naka, Ibaraki
  - 1218.23.15 Boehringer Ingelheim Investigational Site, Nishi-ku, Hiroshima, Hiroshima
  - 1218.23.34 Boehringer Ingelheim Investigational Site, Nishi-ku, Sakai, Osaka
  - 1218.23.22 Boehringer Ingelheim Investigational Site, Nishishinjyuku, Shinjyuku-ku, Tokyo
  - 1218.23.16 Boehringer Ingelheim Investigational Site, Oita, Oita
  - 1218.23.40 Boehringer Ingelheim Investigational Site, Oita, Oita
  - 1218.23.36 Boehringer Ingelheim Investigational Site, Okayama, Okayama
  - 1218.23.11 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1218.23.12 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1218.23.32 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1218.23.33 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1218.23.35 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1218.23.17 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1218.23.18 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1218.23.19 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1218.23.41 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1218.23.42 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1218.23.43 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1218.23.01 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 1218.23.20 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 1218.23.46 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 1218.23.08 Boehringer Ingelheim Investigational Site, Shinjyuku-ku,Tokyo
  - 1218.23.14 Boehringer Ingelheim Investigational Site, Suita, Osaka
  - 1218.23.31 Boehringer Ingelheim Investigational Site, Takatsuki, Osaka
  - 1218.23.48 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa

REFERENCES:
- [Derived] Johansen OE, Neubacher D, von Eynatten M, Patel S, Woerle HJ. Cardiovascular safety with linagliptin in patients with type 2 diabetes mellitus: a pre-specified, prospective, and adjudicated meta-analysis of a phase 3 programme. Cardiovasc Diabetol. 2012 Jan 10;11:3. doi: 10.1186/1475-2840-11-3. PMID 22234149
- [Derived] Horie Y, Hayashi N, Dugi K, Takeuchi M. Design, statistical analysis and sample size calculation of a phase IIb/III study of linagliptin versus voglibose and placebo. Trials. 2009 Sep 5;10:82. doi: 10.1186/1745-6215-10-82. PMID 19732457

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 6 groups (including sub-groups in placebo and voglibose groups)
Pre-assignment Details: Placebo group has 2 sub-groups, placebo-linagliptin 5mg (from 2nd stage) and placebo-linagliptin 10mg (from 2nd stage).
  Both Linagliptin 5 mg and 10 mg groups don't have sub-group. Voglibose group has 2 sub-groups, voglibose-linagliptin 5mg (from 3rd stage) and voglibose-linagliptin 10mg (from 3rd stage).
Groups:
- Placebo - BI1356 (Linagliptin) 5mg - Linagliptin 5mg: Placebo in Stage 1 - 5 mg in Stage 2 - 5 mg in Stage 3
- Placebo - Linagliptin 5mg - Linagliptin 10mg: Placebo in Stage 1 - 10 mg in Stage 2 - 10 mg in Stage 3
- Linagliptin 5mg - Linagliptin 5mg - Linagliptin 5mg: 5 mg in Stage 1 - 5 mg in Stage 2 - 5 mg in Stage 3
- Linagliptin 10 mg - Linagliptin 10 mg - Linagliptin 10 mg: 10 mg in Stage 1 - 10 mg in Stage 2 - 10 mg in Stage 3
- Voglibose - Voglibose - Linagliptin 5mg: Voglibose in Stage 1 - Voglibose in Stage 2 - 5 mg in Stage 3
- Voglibose - Voglibose - Linagliptin 10mg: Voglibose in Stage 1 - Voglibose in Stage 2 - 10 mg in Stage 3
Period: 1st Stage
Arm/Group | Placebo - BI1356 (Linagliptin) 5mg - Linagliptin 5mg | Placebo - Linagliptin 5mg - Linagliptin 10mg | Linagliptin 5mg - Linagliptin 5mg - Linagliptin 5mg | Linagliptin 10 mg - Linagliptin 10 mg - Linagliptin 10 mg | Voglibose - Voglibose - Linagliptin 5mg | Voglibose - Voglibose - Linagliptin 10mg
Started | 39 | 41 | 159 | 160 | 81 | 81
Completed | 36 | 38 | 156 | 155 | 79 | 79
Not Completed | 3 | 3 | 3 | 5 | 2 | 2
Not completed — Adverse Event | 3 | 3 | 3 | 3 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Investigator's decision | 0 | 0 | 0 | 1 | 0 | 0
Period: 2nd Stage
Arm/Group | Placebo - BI1356 (Linagliptin) 5mg - Linagliptin 5mg | Placebo - Linagliptin 5mg - Linagliptin 10mg | Linagliptin 5mg - Linagliptin 5mg - Linagliptin 5mg | Linagliptin 10 mg - Linagliptin 10 mg - Linagliptin 10 mg | Voglibose - Voglibose - Linagliptin 5mg | Voglibose - Voglibose - Linagliptin 10mg
Started | 36 | 38 | 156 | 155 | 79 | 79
Completed | 34 | 38 | 153 | 151 | 71 | 76
Not Completed | 2 | 0 | 3 | 4 | 8 | 3
Not completed — Adverse Event | 2 | 0 | 2 | 3 | 7 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Investigator's decision | 0 | 0 | 1 | 1 | 0 | 0
Period: Extension Stage
Arm/Group | Placebo - BI1356 (Linagliptin) 5mg - Linagliptin 5mg | Placebo - Linagliptin 5mg - Linagliptin 10mg | Linagliptin 5mg - Linagliptin 5mg - Linagliptin 5mg | Linagliptin 10 mg - Linagliptin 10 mg - Linagliptin 10 mg | Voglibose - Voglibose - Linagliptin 5mg | Voglibose - Voglibose - Linagliptin 10mg
Started | 34 | 38 | 153 | 151 | 71 | 76
Completed | 33 | 36 | 142 | 142 | 68 | 73
Not Completed | 1 | 2 | 11 | 9 | 3 | 3
Not completed — Adverse Event | 1 | 2 | 9 | 7 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 1 | 1
Not completed — Closure of the trial site | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: The patients with placebo at the start of randomised study medication
- Linagliptin 5mg: The patients with linagliptin 5 mg at the start of randomised study medication
- Linagliptin 10 mg: The patients with linagliptin 10 mg at the start of randomised study medication
- Voglibose: The patients with voglibose at the start of randomised study medication
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin 5mg | Linagliptin 10 mg | Voglibose | Total
Number analyzed (Participants) | 80 | 159 | 160 | 162 | 561
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (8.9) | 60.3 (9.4) | 61.3 (10) | 58.5 (9.9) | 60.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 48 | 48 | 47 | 166
  Male | 57 | 111 | 112 | 115 | 395

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 12
Description: Change from the baseline measurement, where the baseline measurement was obtained at randomization (0 week) before receiving study medication
Time Frame: 12 weeks
Population: For the 12-week analysis, it was planed the comparison between Linagliptin and placebo. Then the patients with voglibose were excluded in this analysis.Full analysis set for 12-week treatment period with Last Observation Carried Forward.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin 5mg | Linagliptin 10 mg
Number analyzed (Participants) | 80 | 159 | 157
Percent | 0.63 (0.08) | -0.24 (0.06) | -0.25 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5mg; Linagliptin 5 mg vs placebo at week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; Model includes treatment,baseline HbA1c, and number of previous antidiabetic medication; Least Squares Mean Difference = -0.87, 95% CI 2-sided [-1.04 to -0.7], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Placebo vs Linagliptin 10 mg; Linagliptin 10 mg vs placebo at week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; Model includes treatment,baseline HbA1c, and number of previous antidiabetic medication; Least Squares Mean Difference = -0.88, 95% CI 2-sided [-1.05 to -0.71], Standard Error of Mean 0.09

2. Primary Outcome: Change From Baseline in HbA1c at Week 26
Description: as for outcome 1
Time Frame: 26 weeks
Population: For the 26-week analysis, it was planed the comparison between Linagliptin and Voglibose. Then the patients with placebo were excluded in this analysis.Full analysis set for 26-week treatment period with Last Observation Carried Forward.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Linagliptin 5mg | Linagliptin 10 mg | Voglibose
Number analyzed (Participants) | 159 | 157 | 162
Percent | -0.13 (0.07) | -0.19 (0.07) | 0.19 (0.07)
Statistical Analysis 1: Comparison: Linagliptin 5mg vs Voglibose; Test type: Superiority or Other; p = 0.0003, ANCOVA; Model includes treatment,baseline HbA1c, and number of previous antidiabetic medication; Least Squares Mean Difference = -0.32, 95% CI 2-sided [-0.49 to -0.15], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Linagliptin 10 mg vs Voglibose; Linagliptin 10 mg vs voglibose at week 26; Test type: Superiority or Other; p < 0.0001, ANCOVA; Model includes treatment,baseline HbA1c, and number of previous antidiabetic medication; Least Squares Mean Difference = -0.39, 95% CI 2-sided [-0.56 to -0.21], Standard Error of Mean 0.09

3. Secondary Outcome: Relative Efficacy Response of HbA1c at Week 12
Description: HbA1c value decreased below 7.0%, below 6.5% and reduction from baseline ≥0.5% at Week 12
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Linagliptin 5mg | Linagliptin 10 mg
Number analyzed (Participants) | 80 | 159 | 157
Participants
  HbA1c <7.0% | 8 | 42 | 56
  HbA1c <6.5% | 0 | 15 | 18
  HbA1c reduction from baseline ≥0.5% | 7 | 91 | 94

4. Secondary Outcome: Relative Efficacy Response of HbA1c at Week 26
Description: HbA1c value decreased below 7.0%, below 6.5% and reduction from baseline ≥0.5% at Week 26
Time Frame: 26 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Linagliptin 5mg | Linagliptin 10 mg | Voglibose
Number analyzed (Participants) | 159 | 157 | 162
Participants
  HbA1c <7.0% | 48 | 54 | 36
  HbA1c <6.5% | 15 | 21 | 7
  HbA1c reduction from baseline ≥0.5% | 91 | 84 | 61

5. Secondary Outcome: Relative Efficacy Response of HbA1c at Week 52
Description: HbA1c value decreased below 7.0%, below 6.5% and reduction from baseline ≥0.5% at Week 52
Time Frame: 52 weeks
Population: For the 52-week analysis, it was planed to analyse for Linagliptin 5mg and 10mg. Then the patients with placebo and voglibose were excluded in this analysis. Full analysis set for 52-week treatment period with Last Observation Carried Forward
Measure: Number; unit: Participants
Groups:
- Linagliptin 10mg: The patients with linagliptin 10 mg at the start of randomised study medication
Arm/Group | Linagliptin 5mg | Linagliptin 10mg
Number analyzed (Participants) | 159 | 157
Participants
  HbA1c <7.0% | 38 | 29
  HbA1c <6.5% | 6 | 10
  HbA1c reduction from baseline ≥0.5% | 62 | 62

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 12
Description: as for outcome 1
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5mg | Linagliptin 10 mg
Number analyzed (Participants) | 80 | 159 | 160
mg/dL | 7.4 (2.5) | -12.3 (1.9) | -13.0 (1.9)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5mg; Linagliptin 5 mg vs placebo at week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; Model includes treatment,baseline FPG, and number of previous antidiabetic medication; Least Squares Mean Difference = -19.7, 95% CI 2-sided [-25.4 to -14.0], Standard Error of Mean 2.9
Statistical Analysis 2: Comparison: Placebo vs Linagliptin 10 mg; Linagliptin 10 mg vs placebo at week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; Model includes treatment,baseline FPG, and number of previous antidiabetic medication; Least Squares Mean Difference = -20.4, 95% CI 2-sided [-26.2 to -14.7], Standard Error of Mean 2.9

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: as for outcome 1
Time Frame: 26 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Linagliptin 5mg | Linagliptin 10 mg | Voglibose
Number analyzed (Participants) | 159 | 160 | 162
mg/dL | -5.0 (2.4) | -7.8 (2.4) | 2.0 (2.4)
Statistical Analysis 1: Comparison: Linagliptin 5mg vs Voglibose; Linagliptin 5 mg vs Voglibose at week 26; Test type: Superiority or Other; p = 0.0239, ANCOVA; Model includes treatment,baseline FPG, and number of previous antidiabetic medication; Least Squares Mean Difference = -6.9, 95% CI 2-sided [-13.0 to -0.9], Standard Error of Mean 3.1
Statistical Analysis 2: Comparison: Linagliptin 10 mg vs Voglibose; Linagliptin 10 mg vs voglibose at week 26; Test type: Superiority or Other; p = 0.0015, ANCOVA; Model includes treatment,baseline FPG, and number of previous antidiabetic medication; Least Squares Mean Difference = -9.8, 95% CI 2-sided [-15.8 to -3.8], Standard Error of Mean 3.1

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 52
Description: as for outcome 1
Time Frame: 52 weeks
Population: The patients who had at least one available baseline FPG measurement under the treatment with linagliptin
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Linagliptin 5mg | Linagliptin 10 mg
Number analyzed (Participants) | 159 | 160
mg/dL | -3.2 (2.7) | -5.9 (2.7)

9. Primary Outcome: Examination of Long-term Safety of Linagliptin (52-week Treatment)
Description: The incidence of AEs (Preferred Terms) with a frequency of 5% or more in the patients with type 2 diabetes mellitus who received linagliptin (5 mg or 10 mg) once daily for 52 weeks
Time Frame: 52 weeks
Population: The patients who received at least one dose of linagliptin 5 mg or linagliptin 10 mg during the randomised treatment period
Measure: Number; unit: participants
Arm/Group | Linagliptin 5mg | Linagliptin 10 mg
Number analyzed (Participants) | 266 | 274
participants
  Nasopharyngitis | 84 | 81
  Back pain | 15 | 21
  Constipation | 12 | 19

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Placebo (1st Stage) | Linagliptin 5mg (2nd-Extension Stage After Placebo) | Linagliptin 10mg (2nd-Extension Stage After Placebo) | Linagliptin 5mg (1st-2nd-Extension Stage) | Linagliptin 10mg (1st-2nd-Extension Stage) | Voglibose (1st-2nd Stage) | Linagliptin 5mg (Extension Stage After Voglibose) | Linagliptin 10mg (Extension Stage After Voglibose)
Serious Adverse Events (participants affected / at risk) | 1/80 | 3/36 | 1/38 | 14/159 | 10/160 | 7/162 | 3/71 | 3/76
Other Adverse Events (participants affected / at risk) | 23/80 | 19/36 | 21/38 | 101/159 | 107/160 | 83/162 | 28/71 | 31/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (1st Stage) (N=80) | Linagliptin 5mg (2nd-Extension Stage After Placebo) (N=36) | Linagliptin 10mg (2nd-Extension Stage After Placebo) (N=38) | Linagliptin 5mg (1st-2nd-Extension Stage) (N=159) | Linagliptin 10mg (1st-2nd-Extension Stage) (N=160) | Voglibose (1st-2nd Stage) (N=162) | Linagliptin 5mg (Extension Stage After Voglibose) (N=71) | Linagliptin 10mg (Extension Stage After Voglibose) (N=76)
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Limb deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Airway burns (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (1st Stage) (N=80) | Linagliptin 5mg (2nd-Extension Stage After Placebo) (N=36) | Linagliptin 10mg (2nd-Extension Stage After Placebo) (N=38) | Linagliptin 5mg (1st-2nd-Extension Stage) (N=159) | Linagliptin 10mg (1st-2nd-Extension Stage) (N=160) | Voglibose (1st-2nd Stage) (N=162) | Linagliptin 5mg (Extension Stage After Voglibose) (N=71) | Linagliptin 10mg (Extension Stage After Voglibose) (N=76)
Nasopharyngitis (Infections and infestations) | 10 | 10 | 8 | 60 | 57 | 36 | 14 | 16
Rhinitis (Infections and infestations) | 0 | 2 | 2 | 2 | 3 | 2 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 2 | 7 | 6 | 4 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 2 | 3 | 1 | 4 | 1 | 2
Gastroenteritis (Infections and infestations) | 1 | 1 | 2 | 4 | 3 | 2 | 3 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 3 | 0 | 7 | 7 | 7 | 1 | 4
Depression (Psychiatric disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 3 | 2 | 4 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 3 | 2 | 2 | 2 | 2 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 9 | 10 | 2 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 3 | 3 | 2 | 2 | 1
Constipation (Gastrointestinal disorders) | 5 | 0 | 4 | 12 | 12 | 5 | 0 | 3
Dental caries (Gastrointestinal disorders) | 0 | 0 | 2 | 7 | 5 | 4 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 10 | 6 | 15 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 7 | 10 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 6 | 5 | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 4 | 3 | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 11 | 15 | 6 | 1 | 4
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 5 | 4 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.